CLINICAL TRIAL: NCT06644508
Title: The Efficient PICU Fluid Care Evaluation
Acronym: LESSER-2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2023-16717
Record Dates: First submitted 2024-10-10; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-09

CONDITIONS: Respiratory Insufficiency Requiring Mechanical Ventilation; Fluid Overload; Fluid Balance
Keywords: Respiratory Insufficiency; Mechanical ventilation; Fluids; Fluid Balance; Edema; Fluid Overload; Lenght of mechanical ventilation; Childeren; Maintenance fluids
MeSH Terms: conditions — Edema; Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Multicentre prospective study (clinical implementation evaluation) with a before-after design with continuous recruitment and single measurements
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Observation of current local practices (No Intervention): Current local practices regarding fluid management will be observed. Population: Critically ill children receiving mechanical ventilation due to respiratory insufficiency. Patients will be treated according to local protocols at the discretion of the attending physicians.
- Strict adherence to european guidelines (Active Comparator): In this intervention attending physicians will be encouraged to strictly adhere the European (ESPNIC) guidelines regarding fluid management.
  Interventions: Other: Strict adherence to European guidelines

INTERVENTIONS:
Other: Strict adherence to European guidelines — The goal is to maintain a neutral fluid balance throughout the course of intubation if clinical practice allows. Therefore:
  * From the start of mechanical ventilation, the maximum maintenance fluids is 65% of the maintenance fluids proposed by the Holliday & Segar formula. Fluid resuscitation in the first hours after intubation is at the discretion of the attending physician.
  * Any other interventions to maintain a neutral fluid balance (e.g., starting diuretics, reducing fluid boluses, decreasing creep fluids, or using more concentrated enteral feeding) are at the discretion of the attending physician.
  * Throughout the intervention, the attending physician decides if clinical practice allows for a decrease in fluid balance, and international feeding goals must always be met.
  Arms: Strict adherence to european guidelines

SUMMARY:
The goal of this clinical trial is to evaluate and prevent fluid overload in critically ill, mechanically ventilated children. The main questions it aims to answer are:

1. What is the effect of a restrictive fluid strategy on cumulative fluid balance on day three of invasive mechanical ventilation?
2. What is the feasibility (e.g. adherence to target intake, fluid balance and nutritional goals) of maintaining a neutral fluid balance?

Researchers will compare the effects of strict adherence to the European Society of Paediatric and Neonatal Intensive Care (ESPNIC) guidelines regarding fluid balance (i.e. restricting fluid intake and preventing a positive fluid balance) to current local practice.

From the start to the end of invasive mechanical ventilation participants will be treated according to local practice or with the strict aim to prevent a positive fluid balance. Aiming to prevent a positive fluid balance, if this is possible given the clinical context, is at descretion of the attending physician. Minimal caloric intake requirements must be met.

Participants are studied for ten days during invasive mechanical ventilation or until discharge from the intensive care

DETAILED DESCRIPTION:
Objectives

* Compare current practices with strict adherence to ESPNIC guidelines regarding fluid management in critically ill children.
* Assess the effectiveness of maintaining a neutral cumulative fluid balance by day 3 (CFB3).

Study Design

* Type: Multicenter prospective study with a before-after design, continuous recruitment, and single measurements.
* Groups:

  1. Current practice group.
  2. ESPNIC guideline adherence group (restrictive fluid management).

Treatment

* Current Practice Group: Standard PICU treatment per local protocols.
* ESPNIC Guideline Adherence Group: Strict restrictive fluid strategy beginning within 24 hours of intubation, focusing on preventing cumulative positive fluid balance. ESPNIC guidelines recommend restricting total fluid intake to 65-80% of the Holliday and Segar formula. The Holliday and Segar formula is tailored for children under 10 kg: 150 ml/kg/day for neonates and 100 ml/kg/day for one-year-olds. This study will aim for a 65% restriction based on these calculations.

Feeding Enteral nutrition starts within 24-48 hours unless contraindicated, with caloric intake reaching 100% of resting energy expenditure by day 7 and protein intake exceeding 1.5 g/kg/day.

Diuretics The choice and route of diuretics will be at the treating physician's discretion.

Duration of Intervention Start: Onset of mechanical ventilation. End: End of mechanical ventilation.

Study Procedures Children will have routine blood samples taken daily during invasive mechanical ventilation (IMV), which align with standard clinical diagnostics. Body weight will be measured at admission, on day 3, and before extubation. Data on fluid intake, feeding, medication, and urine output will be gathered prospectively in the electronic patient dossier (EPD).

Adverse Events All adverse events will be recorded, with serious adverse events (SAEs) reported to the sponsor promptly.

ELIGIBILITY:
Inclusion Criteria:

* Age < 10 years and weight < 35 kg
* Receiving invasive mechanical ventilation (IMV) due to respiratory failure
* Inclusion possible within 24 hours of start of IMV
* Expected duration of IMV > 48 hours

Exclusion Criteria:

* Preterm (<37weeks gestational age)
* Preexistent (clinical) diagnosis of kidney disease
* Congenital cardiac defect with hemodynamic consequences or reduced cardiac function
* (Ongoing) shock with need for fluid resuscitation and/or vasoactive drugs
* Cardiovascular (including diuretics) drug use on admission (home medication)
* Pre-existent (clinical) diagnosis of liver failure
* Right of left heart failure
* Pulmonary hypertension
* ECMO treatment
* Receiving total parenteral nutrition on admission which won't be stopped
* Failure to include within 12 hours after start of IMV
* Expected duration of IMV < 48 hours
* Parents or caretakers unable to understand/speak Dutch language
* Surgery < 48 hours

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Cumulative fluid balance on day 3 in ml/kg | From start mechanical ventilation to 72 hours after start of mechanical ventilation
  Cumulative fluid balance (CFB) over the course of three days after the start of mechanical ventilation is noted in ml/kg. CFB is calculated as a sum of daily (fluid intake [liters] - total output [liters])/ body weight (kilograms).

SECONDARY OUTCOMES:
Daily cumulative fluid balance on in ml/kg | For 10 days, CFB is noted every day at 00:00
  Daily cumulative fluid balance (CFB) over the course of mechanical ventilation is noted in ml/kg. CFB is calculated as a sum of daily (fluid intake [liters] - total output [liters])/ body weight (kilograms).
Protein intake in gr/kg/day | For ten days after start of mechanical ventilation
  Protein intake in gr/kg/day will be daily noted
Bodyweight in grams | Bodyweight in grams will be measured at start of mechanical ventilation and at 72 hours after start of mechanical ventilation
  Bodyweight in grams
Daily cumulative diuretics dose in mg/kg | From start of mechnical ventilation for ten days, cumulative diuretic dose will be noted at 00:00
  Cumulative diuretics dose will be daily noted in mg/kg.
Blood urea nitrogen (BUN) in mmol/L | BUN will be measured at 24 hours, 72 hours and at 120 hours after start of mechanical ventilation
  During the course of mechanical ventilation blood urea nitrogen (BUN) is measured in mmol/L
Daily creatinine level in µmol/L | Creatinine levels will be noted at: 24, 72 hours and 120 after start of mechanical ventilation
  Daily creatinine level in µmol/L
Daily KDIGO stages (1,2 or 3) will be noted every 24 hours | From start of mechanical ventilation to 120 hours after start of mechanical ventilation.
  Daily KDIGO stages will be noted every 24 hours depending on their urine production. KDIGO 1= <0.5ml/kg/h for 6-12 hours, KDIGO 2 = <0.5ml/kg/h for >12 hours, KDIGO 3 = <0.3ml/kg/h for 24 hours or anuria for >12 hours
Daily potassium levels in mmol/L every 24 hours | From start of mechanical ventilation for ten days, at 08:00 in the morning
  During mechanical ventilation daily potassium levels in mmol/L every 24 hours
Daily sodium levels in mmol/L every 24 hours | From start of mechanical ventilation for ten days, at 08:00 in the morning
  During mechanical ventilation daily sodium levels in mmol/L every 24 hours
Daily lactate measurement in mmol/L every 24 hours | From start of mechanical ventilation for ten days, at 08:00 in the morning
  During mechanical ventilation daily lactate measurement in mmol/L every 24 hours
Daily pH measurement every 24 hours | From start of mechanical ventilation for ten days, at 08:00 in the morning
  During mechanical ventilation daily pH measurement every 24 hours
Daily ketone levels in blood every 24 hours in mmol/L | From start of mechanical ventilation for ten days, at 08:00 in the morning
  During mechanical ventilation daily ketone levels in blood every 24 hours in mmol/L
Daily vasoactive-inotropic score every 24 hours | From start of mechanical ventilation for ten days
  Vasoactive-inotropic score is calculated by: [dopamine dose (μg/kg/min) + dobutamine dose (μg/kg/min) + 100 × epinephrine dose (μg/kg/min) + 10 × milrinone dose (μg/kg/min) + 10 000 × vasopressin dose (unit/kg/min) + 100 × norepinephrine dose (μg/kg/min)]
Daily highest heart rate in beats per minute from every previous 24 hours | From start of mechanical ventilation for ten days
  Daily highest heart rate in beats per minute from every previous 24 hours
Daily lowest heart rate in beats per minute from every previous 24 hours | From start of mechanical ventilation for ten days
  Daily lowest heart rate in beats per minute from every previous 24 hours
Daily mean mean arterial pressure (so mean MAP) over every previous 24 hours | From start of mechanical ventilation for ten days
  Daily mean mean arterial pressure (so mean MAP) over every previous 24 hours. Mean MAP is calculated by calculating the mean from blood pressure from hourly collected data
Daily mean heart rate in beats per minute over every previous 24 hours | From start of mechanical ventilation for ten days
  Daily mean heart rate in beats per minute over every previous 24 hours. Mean Mean heart rate is calculated by calculating the mean heartrate from hourly collected data
Duration of IMV in days | From start of mechanical ventilation for ten days
  Duration of invasive mechanical ventilation is noted in days
Duration of high flow nasal canula therapy after end of mechanical ventilation in hours | From the end of mechanical ventilation up to ten days after start of mechanical ventilation
  Duration of high flow nasal canula therapy after end of mechanical ventilation in hours
Need for extracorporeal organ support (ECMO) is noted (yes/no) | From start of mechanical ventilation to day ten after start of emchanical ventilation
  Need for extracorporeal organ support (ECMO) is noted (yes/no)
Daily mean oxygenation saturation index is noted every 24 hours only when SpO2 was below 97% | From start of mechanical ventilation for ten days
  During IMV daily mean oxygenation saturation index is noted every 24 hours only when SpO2 was below 97%. This is calculated by: ([Paw x FiO2]/SpO2) × 100
Mean daily P/F ration is noted from every previous 24 hours | From start of mechanical ventilation for ten days
  During IMV mean daily P/F ration is noted from every previous 24 hours
Lenght of pediatric intensive care (PICU) stay in days | From start of mechanical ventilation to 10 days after start mechanical ventilation
  Lenght of pediatric intensive care (PICU) stay in days
Newly acquired pulmonary infections (yes/no) | From start of mechanical ventilation for ten days
  Newly acquired pulmonary infections (yes/no)
Total daily fluid balance is noted in ml/kg every 24 hours | From start of mechnical ventilation for ten dys
  Total daily fluid balance is noted in ml/kg every 24 hours
Daily fluid intake in ml/kg every 24 hours | From start of mechanical ventilation for ten days
  Daily fluid intake will be noted in ml/kg ervery 24 hours
Caloric intake in kcal/kg every 24 hours | From start of mechanical ventilation for ten days
  Daily caloric intake in kcal/kg will be noted every 24 hours
Daily urine production in ml//kg from every 24 hours | From start of mechnical ventilation for ten days
  Daily urine production in ml//kg from every 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Joris Lemson, MD PhD, Principal Investigator — Radboud University Medical Center
Locations (3):
- Netherlands (3):
  - Radboudumc, Nijmegen, Gelderland
  - Amsterdam MC, Amsterdam, North Holland
  - ErasmusMC, Rotterdam, South Holland

IPD SHARING:
Plan to Share IPD: Yes
* Demograpghics data
  * Outcome data
Supporting Information: Study Protocol
Time Frame: From publication until 15 years after publication
Access Criteria: Data will be made available upon reasonable request to the corresponding author

REFERENCES:
- [Background] Arrahmani I, Ingelse SA, van Woensel JBM, Bem RA, Lemson J. Current Practice of Fluid Maintenance and Replacement Therapy in Mechanically Ventilated Critically Ill Children: A European Survey. Front Pediatr. 2022 Feb 23;10:828637. doi: 10.3389/fped.2022.828637. eCollection 2022. PMID 35281243
- [Background] Valentine SL, Sapru A, Higgerson RA, Spinella PC, Flori HR, Graham DA, Brett M, Convery M, Christie LM, Karamessinis L, Randolph AG; Pediatric Acute Lung Injury and Sepsis Investigator's (PALISI) Network; Acute Respiratory Distress Syndrome Clinical Research Network (ARDSNet). Fluid balance in critically ill children with acute lung injury. Crit Care Med. 2012 Oct;40(10):2883-9. doi: 10.1097/CCM.0b013e31825bc54d. PMID 22824936
- [Background] Ingelse SA, Geukers VG, Dijsselhof ME, Lemson J, Bem RA, van Woensel JB. Less Is More?-A Feasibility Study of Fluid Strategy in Critically Ill Children With Acute Respiratory Tract Infection. Front Pediatr. 2019 Dec 10;7:496. doi: 10.3389/fped.2019.00496. eCollection 2019. PMID 31921715
- [Background] Diaz F, Nunez MJ, Pino P, Erranz B, Cruces P. Implementation of preemptive fluid strategy as a bundle to prevent fluid overload in children with acute respiratory distress syndrome and sepsis. BMC Pediatr. 2018 Jun 26;18(1):207. doi: 10.1186/s12887-018-1188-6. PMID 29945586
- [Background] Charaya S, Angurana SK, Nallasamy K, Jayashree M. Restricted versus Usual/Liberal Maintenance Fluid Strategy in Mechanically Ventilated Children: An Open-Label Randomized Trial (ReLiSCh Trial). Indian J Pediatr. 2025 Jan;92(1):7-14. doi: 10.1007/s12098-023-04867-4. Epub 2023 Oct 18. PMID 37851328
- [Background] Brossier DW, Tume LN, Briant AR, Jotterand Chaparro C, Moullet C, Rooze S, Verbruggen SCAT, Marino LV, Alsohime F, Beldjilali S, Chiusolo F, Costa L, Didier C, Ilia S, Joram NL, Kneyber MCJ, Kuhlwein E, Lopez J, Lopez-Herce J, Mayberry HF, Mehmeti F, Mierzewska-Schmidt M, Minambres Rodriguez M, Morice C, Pappachan JV, Porcheret F, Reis Boto L, Schlapbach LJ, Tekguc H, Tziouvas K, Parienti JJ, Goyer I, Valla FV; Metabolism Endocrinology and Nutrition section of the European Society of Pediatric and Neonatal Intensive Care (ESPNIC). ESPNIC clinical practice guidelines: intravenous maintenance fluid therapy in acute and critically ill children- a systematic review and meta-analysis. Intensive Care Med. 2022 Dec;48(12):1691-1708. doi: 10.1007/s00134-022-06882-z. Epub 2022 Oct 26. PMID 36289081